CLINICAL TRIAL: NCT06931119
Title: Aprepitant in the Management of Immune Checkpoint Inhibitors Pruritus: Pilot Study in Solid Cancer Patients
Brief Title: Aprepitant in the Management of Immune Checkpoint Inhibitors Pruritus in Solid Cancer Patients
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Gal Markel, Director Davidoff cancer center, Deputy CEO Rabin medical center, Rabin Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0173-25-RMC
Record Dates: First submitted 2025-04-01; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Pruritus
Keywords: pruritus, immune checkpoint inhibitors
MeSH Terms: conditions — Pruritus | interventions — Aprepitant; Capsules

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- 1 cycle of EMEND® capsules administration (Experimental): 1 cycle (1 administration of EMEND® capsules)
  * Frequency: Patients will take EMEND® capsules at the start of new ICI.
  * Dosing Schedule:
    * Day 1: EMEND® 125 mg, taken orally 1-2 hours before ICI administration.
    * Day 2: EMEND® 80 mg, taken orally in the morning.
    * Day 3: EMEND® 80 mg, taken orally in the morning 7 days after the first capsule of Aprepitant- 12-PSS, safety assessment, QLQ-C30 Follow-up 2- 12-PSS, safety assessment Follow-up 3- 12-PSS, safety assessment Follow-up 4- 12-PSS, QLQ-C30, safety assessment, review of rescue medication use Extended Follow-up- Recurrence of pruritus, long-term safety monitoring, QLQ-C30
  Interventions: Drug: EMEND® (EE mend) (aprepitant) capsules (80mg +125mg) Marketing Authorization Holder and Importer: Merck Sharp & Dohme (Israel-1996) Company Ltd.

INTERVENTIONS:
Drug: EMEND® (EE mend) (aprepitant) capsules (80mg +125mg) Marketing Authorization Holder and Importer: Merck Sharp & Dohme (Israel-1996) Company Ltd. — Total Treatment Duration: 1 cycle (1 administration of EMEND® capsules)
  * Frequency: Patients will take EMEND® capsules at the start of new ICI.
  * Dosing Schedule:
    * Day 1: EMEND® 125 mg, taken orally 1-2 hours before ICI administration.
    * Day 2: EMEND® 80 mg, taken orally in the morning.
    * Day 3: EMEND® 80 mg, taken orally in the morning. During the study period (12 weeks), participant must refrain from using any medications that could potentially interfere with the study's assessment of pruritus symptoms (e.g steroids, antihistamines)
  Follow-up 1(7 days after the first capsule of Aprepitant): 12-PSS, safety assessment, QLQ-C30 Follow-up 2: 12-PSS, safety assessment Follow-up 3: 12-PSS, safety assessment Follow-up 4: 12-PSS, QLQ-C30, safety assessment Extended Follow-up: Recurrence of pruritus, long-term safety monitoring, QLQ-C30

SUMMARY:
Pruritus, commonly known as itching, is an unpleasant sensation that triggers the urge to scratch, which may provide temporary relief. Pruritus can be intermittent or persistent, localized or widespread, and may be associated with medication use. Chronic pruritus, defined as lasting more than six weeks, can significantly affect sleep and quality of life.

Dermatologic toxicities are among the most common immune-related adverse events (irAEs), reported in 43-45% of patients receiving ipilimumab and approximately 34% of those treated with nivolumab or pembrolizumab. Combination therapies (ipilimumab+ nivolumab or pembrolizumab) tend to elevate the incidence of potential irAEs to 41%. These toxicities typically emerge within the first few weeks of treatment, though delayed-onset cases have been documented. Cutaneous irAEs occur more rapidly in patients receiving combination therapy compared to anti-PD1 monotherapy.

Pruritus is one of the most frequently observed cutaneous irAEs. Current treatments for pruritus are often inadequate, leaving many patients suffering from persistent and debilitating symptoms. Despite available therapies, a significant number of individuals continue to experience chronic itch that negatively impacts their quality of life. Substance P (SP) functions as a neurotransmitter and neuromodulator in the central and peripheral nervous systems of mammals. It is produced by both neuronal and non-neuronal cells and plays a role in various physiological responses, including nausea, depression, vomiting, pain, neurogenic inflammation, and, more recently, pruritus. SP exerts its biological effects primarily through neurokinin receptors (NKRs), also known as tachykinin receptors. When SP binds to NK1R in the skin, it triggers mast cell degranulation, leading to the release of pruritogenic and proinflammatory mediators such as histamine, interferon-γ, leukotriene B4, vascular endothelial growth factor (VEGF), and nerve growth factor (NGF). This results in vasodilation and neurogenic inflammation, manifesting clinically as pruritus, erythema, and edema. NK1R antagonists are a class of drugs with antiemetic, antidepressant, anxiolytic, and antipruritic properties, though they have not been effective as analgesics in humans. These drugs act centrally by crossing the blood-brain barrier and selectively blocking NK1R activation by SP in the central nervous system, particularly in vomiting centers. Aprepitant has also demonstrated efficacy in treating pruritus induced by anticancer therapies.

This study is a pilot, single-center open label study evaluating the safety and efficacy of single course of EMEND® (aprepitant) capsules (80mg +125mg) in treating pruritus (new onset and/or refractory) induced by immune checkpoint inhibitors in patients with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Histologically confirmed solid tumor (e.g., melanoma, RCC, NSCLC).
* Currently receiving ICIs (such as but not limited to nivolumab, pembrolizumab, ipilimumab)
* Pruritus that is either:
* Refractory: Persistent pruritus despite standard treatment (e.g., antihistamines, corticosteroids).
* New-onset: Developing after initiation of ICIs or targeted therapies.
* ECOG performance status 0-2.
* Willingness to comply with study procedures and provide informed consent.

Exclusion Criteria:

* History of severe allergic reactions to Aprepitant.
* Uncontrolled or severe dermatologic conditions unrelated to cancer therapy.
* Use of NK1R antagonists within 4 weeks before study entry.
* Concurrent use of medications that strongly interact with Aprepitant.
* Concurrent use of medications that may influence pruritus manifestation (e.g steroids or antihistamines) . Note, Regular treatment with such medications prior to the appearance of pruritus, and or pruritus appearing despite such regular treatment, will not disqualify you from participating in the study
* Uncontrolled infection or significant comorbidities.
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-30 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Response is defined as 6 points reduction of pruritus intensity compared to the baseline value. | 12-Item Pruritus Severity Scale (12-PSS) score over a 12 weeks period, at baseline, every 7 days periprocedural for 4 weeks, and up to 12 weeks
  score interpretation: mild (3-6), moderate (7-11), or severe (12-22). higher scores indicate severe pruritus.

SECONDARY OUTCOMES:
Duration of pruritus relieving: the time from pruritus effective relief to 12-PSS score increase | baseline and up to 12 weeks post treatment

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the results publication